CLINICAL TRIAL: NCT05920590
Title: The Effect of Proprioceptive Neuromuscular Facilitation and Tendon Vibration After Total Knee Arthroplasty: A Randomized Clinical Trial
Brief Title: The Effect of Proprioceptive Neuromuscular Facilitation and Tendon Vibration After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Dimitrios Lytras PT, PhD, Senior Lecturer of Physiotherapy, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-09/2023
Record Dates: First submitted 2023-06-17; First posted 2023-06-27 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Knee Osteoarthritis; Total Knee Arthroplastry
Keywords: Knee Osteoarthritis; Total knee arthroplasty; Proprioceptive Neuromuscular Facilitation; Focal Tendon Vibration; Physiotherapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: In this study, 90 patients with knee osteoarthritis scheduled for unilateral total knee arthroplasty will participate. Each will follow a 4-week physiotherapy program immediately after surgery, according to the latest guidelines. The program will start on the second postoperative day in the hospital and continue with home visits after discharge. After the initial 4-week period, participants will be randomly assigned to one of three groups. The first group will follow a six-week PNF exercise protocol (PNF group). The second group will follow the same PNF regimen with added targeted vibration therapy on the tendon of the vastus medialis and rectus femoris (PNF + Tendon Vibration group). The third group (control group) will receive instructions and an exercise leaflet for home practice without additional treatment. The intervention will last six weeks, starting four weeks post-surgery, with measurements at baseline, at the 6th week, and at six months post-intervention.
Who Masked: Outcomes Assessor
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNF Group (Experimental): Participants allocated to this group will receive 18 sessions of therapeutic exercise program based on the PNF concept (Bello et al. 2011).
  Interventions: Other: PNF
- PNF and Tendon Vibration Group (Experimental): Participants allocated to this group will receive the same PNF protocol with Group 1 in combination with the application of tendon vibration.
  Interventions: Other: PNF plus Tendon Vibration
- Control (Active Comparator): Participants allocated to this group will be given an exercise leaflet for home-based exercises
  Interventions: Other: Control

INTERVENTIONS:
Other: PNF — The protocol will be individualized and will last 45 minutes. The following techniques will be applied:
  * Application of the "hold - relax" technique to increase the range of motion of knee flexion.
  * Rhythmic initiation with the application of diagonal trunk and lower limb shapes.
  * Application of stabilizing reversals from a sitting and standing position.
  * Application of dynamic reversals from a standing position.
  * Rhythmic stabilization.
  * Combination of isotonics.
  * Gait retraining.
  Arms: PNF Group
Other: PNF plus Tendon Vibration — Participants in this group will be given the same exercise program as Group 1 combined with the application of tendon vibration. Tendon vibration will be applied on both quadriceps' tendons in three weekly sessions (not on the same day as the exercise program). To implement the protocol, 100 Hz frequency mechanical stimulation will be applied.
  Arms: PNF and Tendon Vibration Group
Other: Control — Participants in this group will be given an exercise leaflet for home-based exercises and will be instructed to perform these exercises three times a week for the same period as the other two groups (6 weeks). They will also be given recommendations to maintain and increase their physical activity.
  Arms: Control

SUMMARY:
Knee osteoarthritis is a degenerative joint disease characterized by the destruction and progressive loss of articular cartilage. In an advanced stage of the disease, the patient undergoes a total knee joint replacement with an artificial joint (total arthroplasty). The aim of this clinical study is to investigate the effect of combining a therapeutic exercise program based on Proprioceptive Neuromuscular Facilitation (PNF) and tendon vibration in older adult patients after total knee arthroplasty (TKA). Ninety (90) adults over 65 years of age who will undergo TKA due to knee osteoarthritis will be divided into three groups of 30 people each (two intervention and one control). The participants in the first group will follow a therapeutic exercise protocol based on the PNF technique for six weeks. The participants in the second intervention group will follow the same therapeutic exercise program based on PNF, and at the same time, tendon vibration will be applied on the common insertion tendon of the rectus femoris and vastus medialis for the same period. Finally, the participants in the third group (control group) will receive instructions for performing exercises at home via a leaflet without receiving any additional treatment. The subjective perception of pain with the Numeric Pain Rating Scale (NPRS), active range of motion (AROM) of knee flexion with a goniometer, functional ability with the Knee Injury and Osteoarthritis Outcome Score (KOOS), quality of life with the Western Ontario and McMaster Universities Arthritis Index (WOMAC), balance using the Timed Up and Go (TUG) test and Berg Balance Scale (BBS), center of mass displacement with a force platform, and knee proprioception through the calculation of joint position sense using the joint repositioning test will be assessed at the beginning of the intervention (4 weeks post-surgery), at the 6th week, and six months post-intervention. For the statistical analysis of the results, a two-factor analysis of variance with repeated measurements will be applied, with the statistical significance level set at p < .05.

DETAILED DESCRIPTION:
Background: Knee osteoarthritis is a degenerative joint disease characterized by destruction and progressive loss of articular cartilage. It occurs more often in older adults and is accompanied by pain, stiffness and swelling of the knee joint, difficulty in walking, and a decrease in the functioning of the patient. In an advanced stage of the disease, the patient undergoes a total replacement of the knee joint with an artificial joint (total arthroplasty).

Aim: The aim of this clinical study is to investigate the effect of combining a therapeutic exercise program based on Proprioceptive Neuromuscular Facilitation (PNF) and tendon vibration in older adult patients after total knee arthroplasty (TKA).

Method: Ninety (90) adults over 65 years of age who will undergo TKA due to knee osteoarthritis will be divided into three groups of 30 people each (two intervention and one control). The participants in the first group will follow a therapeutic exercise protocol based on the PNF technique for six weeks. The participants in the second intervention group will follow the same therapeutic exercise program based on PNF, and at the same time, tendon vibration will be applied on the common insertion tendon of the rectus femoris and vastus medialis for the same period. Finally, the participants in the third group (control group) will receive instructions for performing exercises at home via a leaflet without receiving any additional treatment. The subjective perception of pain with the Numeric Pain Rating Scale (NPRS), active range of motion (AROM) of knee flexion with a goniometer, functional ability with the Knee Injury and Osteoarthritis Outcome Score (KOOS), quality of life with the Western Ontario and McMaster Universities Arthritis Index (WOMAC), balance using the Timed Up and Go (TUG) test and Berg Balance Scale (BBS), center of mass displacement with a force platform, and knee proprioception through the calculation of joint position sense using the joint repositioning test will be assessed at the beginning of the intervention (4 weeks post-surgery), at the 6th week, and six months post-intervention. For the statistical analysis of the results, a two-factor analysis of variance with repeated measurements will be applied, with the statistical significance level set at p < .05.

Expected results: It is known that older adults with TKA present deficits in balance and knee proprioception due to the long-term functional limitations caused by the symptoms of the disease (difficulty and pain during standing and movement, impaired gait patterns). These deficits persist even after TKA, making older adults more vulnerable to falls and future injuries. Both PNF and tendon vibration are effective therapeutic approaches for proprioception training in older adults. The investigators believe that the inclusion of tendon vibration in the PNF-based therapeutic exercise program will further increase the balance and proprioceptive ability of older adults, while at the same time accelerating their recovery process. Additionally, the effectiveness of an exercise program based on PNF has not been sufficiently studied.

ELIGIBILITY:
Inclusion Criteria:

* Age over 65 years
* Unilateral primary total knee arthroplasty
* Body mass index less than 30
* Active knee flexion range of motion of at least 90° two weeks after surgery
* Written consent to participate in the research

Exclusion Criteria:

* Non-ambulatory patients with knee osteoarthritis
* Infections and other surgical complications following the procedure that result in prolonged hospitalization
* Neurodegenerative disease (e.g., Parkinson's)
* Cognitive deficits - dementia (Mini Mental State Exam Test score < 23)

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
Changes in neck pain intensity with Numeric Pain Rating Scale (NPRS) | pre-treatment, week 6, 6-month follow-up
  This tool is an eleven-point pain scale numbered from zero to 10. The left end of the scale corresponds to zero and is marked as "No pain", whereas the right end corresponds to 10 and is marked as "Maximum pain". Consequently, a higher value indicates more intense pain (Childs et al, 2005). The examinee is asked to choose an integer that best reflects the intensity of their pain. The NPRS is widely used to measure pain in both clinical practice and research, showing high test-retest reliability and high conceptual construct validity.
Changes in active Range of Motion (active ROM) of the knee joint flexion | pre-treatment, week 6, 6-month follow-up
  Active range of knee flexion will be assessed with a long arm goniometer. The measurement will be performed with the subject supine on the examination bed based on the instructions by Hancock et al. (2018), according to whom, measurement with a long arm goniometer shows very high reliability. Three consecutive bends will be requested from the examinee and the highest measured value will be recorded.
3. Changes in functional capacity with the Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire | pre-treatment, week 6, 6-month follow-up
  The KOOS questionnaire is a self-report tool for assessing functional limitations related to knee injuries or osteoarthritis (Roos et al., 1998). It is used in both research to assess functional ability and in clinical practice. The questionnaire includes 42 questions divided into five subscales: knee pain (KOOS pain), other knee symptoms (KOOS symptoms), functional limitations (KOOS ADL), ability to participate in sports or leisure activities (KOOS Sport/Rec), and quality of life (KOOS QOL). A five-point Likert scale from 0 (No problems) to 4 (Extreme problems) is used to score the questionnaire. Each of the KOOS subscales is scored separately, representing different aspects of the functional limitations experienced by the patient. The score for each subscale is converted to a 100-point scale, where a higher score indicates fewer functional limitations.
Changes in quality of life with Western Ontario and McMaster Universities Arthritis (WOMAC) index | pre-treatment, week 6, 6-month follow-up
  The WOMAC index is widely used in the assessment of the quality of life of people with osteoarthritis of the hip and knee (Salafi et al. 2005). It is a self-report questionnaire consisting of 24 questions classified into three subscales: Pain, knee joint stiffness and functional ability in everyday skills.Test questions are scored on a scale of 0 to 4. Scores for each subscale are summed, with a possible score range of 0-20 for pain, 0-8 for stiffness, and 0-68 for functional ability. A sum of the scores for all three subscales gives a total WOMAC score. The higher the score, the less functional the joint.The internal consistency of the subcategories of the Greek WOMAC version ranges from high (0.804) to excellent (0.956), while the intra-class correlation coefficients for test-retest reliability have been characterized as excellent (ranging between 0.91 - 0.95) (Papathanasiou et al. 2015).
Changes in Timed Up and Go test | pre-treatment, week 6, 6-month follow-up
  It is a simple test used to assess a person's mobility. It requires both static and dynamic balance and is a valid and reliable indicator of the functional ability of an individual (Podsiadlo & Richardson, 1991). The participant starts in a seated position. They then stand up following the instructions of the therapist, walk three meters, turn around, walk back to the chair and sit down. The examiner tracks time using a stopwatch. Time is calculated in seconds. A higher score indicates lower functional ability of the participant. The TUG shows high reliability indices in older adults both in measurements by different examiners and in measurements by the same examiner at different times (Cameron and Monroe, 2007).
Changes in Berg Balance scale Test | pre-treatment, week: 3, 6, 6-month follow-up
  The Berg Balance Scale is a tool proposed by Berg (Berg et al., 1989; Berg et al., 1992) for assessing balance in the elderly. The test involves the execution of 14 tests of gradual increasing difficulty where in each one, the subject is asked to maintain a given position for a specific time or conduct specific tasks. Each of the 14 tests on the list is graded according to the balancing ability of the examinee from 0 to 4 points (with 0 indicating low balance ability, while 4 indicates high balance ability). According to Berg et al. (1992), a score of 56 indicates functional balance, whereas a score lower than 45 indicates notable balance deficits that have been related to increased fall risk. Studies have shown high intra-rater and inter-rater reliability in the elderly populations with intraclass correlation (ICC) ranging from .98 to .88 (Berg et al. 1992) and high content validity (Telenius et al., 2015).
Changes of center of mass (COM) displacement | pre-treatment, week 6, 6-month follow-up
  Changes in COM displacement will be recorded using static posturography based on the protocol of Brech et al. (2022). Participants will remain barefoot and static for one minute while standing at ease on the force platform with feet shoulder-width apart, gazing at a target placed 2 meters away. Three attempts will be performed with one-minute intervals in between. The same procedure will be repeated with eyes closed. Parameters for measuring static balance under both conditions (eyes open and eyes closed) will include the root mean square of the displacement from the center of pressure (COP) in the mediolateral and anteroposterior directions. Additionally, the maximum range of COP displacement (sum of maximum and minimum displacement/amplitude) in these directions, and the mean velocity from the total COP displacement in all directions will be considered. For calculating the COP displacement area, values representing 95% of the total displacement ellipse will be used.
Chances in knee joint position sense | pre-treatment, week 6, 6-month follow-up
  Joint position sense will be calculated using the repositioning knee joint test according to the protocol of Relph and Herrington (2015). The joint position sense will be evaluated at two angles: 30° and 60°, with the knee moving from full extension (180°) to 90° flexion and vice versa. For the target angles, the participant will be required to replicate the specified angles.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physiotherapy, Faculty of Health Sciences International Hellenic Universit, Thessaloniki, Sindos Thessaloníki, Greece

IPD SHARING:
Plan to Share IPD: No